CLINICAL TRIAL: NCT06301880
Title: Effect of Topically-applied Milrinone or Nitroglycerin on Internal Mammary Artery Free Flow
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Mohammad Bashar Izzat, Professor, Damascus University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3200
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Internal Mammary Artery Syndrome; Vasodilation
Keywords: milrinone; graft; coronary artery bypass grafting; spasm
MeSH Terms: conditions — Aneurysm; Spasm | interventions — Milrinone; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All surgical procedures and measurements were carried out by a single surgeon (MBI) who was blinded to the topical agent which was applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Normal saline (Placebo Comparator): Patients in this group were randomly assigned to receive the topical application of normal saline (0.9% sodium chloride solution) on the LIMA graft as control
  Interventions: Drug: The topical application of a vasodilator on the LIMA graft
- Group 2: Nitroglycerin (Active Comparator): Patients were randomly assigned to receive the topical application of nitroglycerin (Caspian Tamin Pharmaceutical, Guilan, Iran) 10 mg in 20 ml of normal saline on the LIMA graft.
  Interventions: Drug: The topical application of a vasodilator on the LIMA graft
- Group 3: milrinone (Active Comparator): Patients were randomly assigned to receive the topical application of milrinone (Baxter Pharmaceuticals, Ahmedabad, India) on the LIMA graft
  Interventions: Drug: The topical application of a vasodilator on the LIMA graft

INTERVENTIONS:
Drug: The topical application of a vasodilator on the LIMA graft — Patients were randomly assigned to receive the topical application of one of three agents: milrinone (Baxter Pharmaceuticals, Ahmedabad, India) 10 mg in 20 ml of dextrose 5%, nitroglycerin (Caspian Tamin Pharmaceutical, Guilan, Iran) 10 mg in 20 ml of normal saline, or normal saline (0.9% sodium chloride solution) as control.
  Other Names: milrinone (Baxter Pharmaceuticals, Ahmedabad, India), nitroglycerin (Caspian Tamin Pharmaceutical, Guilan, Iran)

SUMMARY:
Forty-six consecutive patients undergoing elective primary coronary artery bypass grafting were enrolled. After the left IMA was harvested, free flow was measured under controlled hemodynamic conditions before any intervention (flow 1) and at a mean of 12.5 minutes after the topical application of one of three agents (milrinone, nitroglycerin or normal saline) on the IMA (flow 2).

DETAILED DESCRIPTION:
Fifty consecutive patients undergoing elective primary coronary artery bypass grafting were enrolled in this study. Patients were randomly assigned to receive the topical application of one of three agents: milrinone (Baxter Pharmaceuticals, Ahmedabad, India) 10 mg in 20 ml of dextrose 5%, nitroglycerin (Caspian Tamin Pharmaceutical, Guilan, Iran) 10 mg in 20 ml of normal saline, or normal saline (0.9% sodium chloride solution) as control.

All surgical procedures and measurements were carried out by a single surgeon who was blinded to the topical agent which was applied. Each patient enrolled in the study gave a written informed consent, and the study protocol conforms to the ethical guidelines of the 1975 Declaration of Helsinki as reflected in a priori approval by the local human research committee.

Operative Technique After sternal incision, the skeletonized left IMA was harvested from the subclavian artery to its bifurcation with low-powered electrocautery, and major collaterals were ligated with hemoclips. Following systemic heparinization (300 units/kg to achieve an activated clotting time target of 480 seconds), the IMA was divided proximal to its bifurcation. The first IMA flow (flow 1) was measured by reading the volume of blood ejected from the tip of the freely bleeding IMA through a one-minute period. Heart rate, mean arterial pressure and central venous pressure were documented at the same time. The tip of the artery was occluded with a bulldog clamp, and a swab which was soaked with the selected vasodilator at room temperature (18.0 to 20.0 degrees C) was wrapped around the IMA, and was left undisturbed until the second set of measurements.

Cannulation for cardiopulmonary bypass was carried out, and the pump was used to transfuse or drain blood from the patient in order to restore the mean arterial and central venous pressures as nearly as possible to the previous values. Systemic vasopressors or vasodilators were not used. The IMA was then unwrapped and the second IMA flow (flow 2) was measured in the same way. Time, heart rate, and mean arterial and central venous pressures were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective primary coronary artery bypass grafting

Exclusion Criteria:

* patients who developed ischemic events during surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
LIMA free flow | Immediately following harvesting the LIMA and 10 mintues following the topical application of the drug
  Reading the volume of blood ejected from the tip of the freely bleeding IMA through a one-minute period

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Bashar Izzat, FRCS(CTh), Principal Investigator — Damascus University
Locations (1):
- Damascus University Cardiac Surgery Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Yes
Data has been deposited in data repository 10.6084/m9.figshare.24905154 License CC BY 4.0
Supporting Information: CSR
Time Frame: Data is currently and permanently available
Access Criteria: open access